CLINICAL TRIAL: NCT04226066
Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability and Pharmacokinetics Characteristics of Recombinant Oncolytic Vaccinia Virus Injection T601 as a Single Drug or in Combination With Oral Flucytosine (5-FC), in Patients With Advanced Malignant Solid Tumors
Brief Title: Safety, Tolerability and Pharmacokinetics Characteristics of Recombinant Oncolytic Vaccinia Virus Injection T601 as a Single Drug or in Combination With Oral Flucytosine (5-FC), in Patients With Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tasly Tianjin Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: T60101
Record Dates: First submitted 2019-12-05; First posted 2020-01-13 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: Advanced Malignant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T601/T601+5-FC (Experimental): Part 1: Dose-escalation study of T601 single-dose; Part 2: Dose-escalation study of T601 single-dose combined with 5-FC; Part 3: Dose-escalation study of T601 multiple-dose combined with 5-FC; Part 4: Extended study of T601 multiple-dose combined with 5-FC.
  Interventions: Biological: T601; Combination Product: T601+5-FC

INTERVENTIONS:
Biological: T601 — Part1: T601 is injected once (Day1). Dose range: 1E+7, 3E+7, 1E+8, 3E+8, 1E+9pfu.Trial cycle: Day1-21.
  For part1, 3+3 dose-escalation. After all patients of one dosage finished DLT evaluation, investigator judged that patients can benefit from treatment and no intolerable toxicity occurred, patients could receive maintenance treatment, and treatment plan is same as Cycle 1.
Combination Product: T601+5-FC — Part2: T601 is injected once (Day1). Dose range: MTD-2, MTD-1 and MTD of Part1. 5-FC is taken on Day5-18 for 14 consecutive days. Trial cycle: Day1-28.
  Part3: T601 is injected 3 times (Day1, 8, 15). Dose range: MTD-1 and MTD, or MTD-2 and MTD-1 of Part2. 5-FC is taken on Day5-7, Day12-14 and Day19-32. Trial cycle: Day1-46.
  Part4: Protocol revised based on results of Part1-Part3. Preliminary plan: 30 patients with gastric cancer, pancreatic cancer and hepatocellular cancer who have failed standard therapeutic options are enrolled (10 patients for each indication). Treatment plan is same as Part3.
  For part2 and part3, 3+3 dose-escalation. After all patients of one dosage finished DLT evaluation, investigator judged that patients can benefit from treatment and no intolerable toxicity occurred, patients could receive maintenance treatment, and treatment plan is same as Cycle 1.

SUMMARY:
This open, dose-escalation and extended PhI/IIa clinical trial aims to evaluate the safety, tolerability of T601 as a single-agent as well as combined with prodrug 5-FC to treat patients with advanced malignant solid tumors and to explore the pharmacokinetic characteristics of T601, 5-FC, 5-FU, FBAL, which includes PhI study of dose-escalation study and Ph IIa study of extending study.

DETAILED DESCRIPTION:
Preclinical studies have confirmed that the combination of T601 and 5-FC can not only enhance the anti-tumor effect, but also reduce the toxicity of T601. Considering the risks and benefits of participants of the clinical trial, the protocol design is divided into 4 parts:

Part 1: dose-escalation study of single-dose of T601 to evaluate the safety and tolerability of T601 and to determine the MTD;

Part 2: dose-escalation study of single-dose of T601 combined with predrug 5-FC, to evaluate the safety and tolerability of the treatment of single dose of T601 combined with predrug 5-FC and to determine the MTD of single dose of T601 when combing with 5-FC;

Part 3: dose-escalation study of multiple-dose of T601 combined with predrug 5-FC, to explore the safety and tolerability of the treatment of multiple dose of T601 combined with predrug 5-FC and to determine the MTD of multiple dose of T601 when combing with 5-FC, also to determine the RP2D (recommended dose for Phase II Trial);

Part 4: extending study of multiple-dose of T601 combined with predrug 5-FC, to evaluate the efficacy of the treatment of multiple-dose of T601 combined with predrug 5-FC in patients with various specific tumors and to evaluate the ORR, DCR and PFS according to the RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years and ≤ 75;
2. Part1-Part3: histological or cytological confirmed advanced malignant solid tumors patients who have received standard therapeutic options in previous treatment and now there's no standard therapy available; Part4: patients with gastric cancer, pancreatic cancer and hepatocellular carcinoma will be enrolled in Phase IIa Clinical Trial;
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
4. Expected survival of at least 3 months;
5. Patient presenting with at least one evaluable lesion according to RECIST 1.1 in Part1-Part3; patient presenting with at least one measurable lesion according to RECIST 1.1 in Part4;
6. Adequate blood system function, liver function and kidney function:

   1. ANC≥1.5×109/L，PLT≥80×109/L，Hb≥90 g/L;
   2. TBIL≤1.5×ULN，ALT≤3×ULN，AST≤3×ULN (Patients with liver metastasis or liver cancer ALT≤5×ULN，AST≤5×ULN);
   3. Cr≤1.5×ULN, creatinine clearance>50mL/min (calculate according to Cockcroft-Gault Formula);
   4. APTT≤1.5×ULN，PT≤1.5×ULN，INR≤1.5×ULN.
7. Fertile eligible patients (male and female) must agree to use highly effective method of contraception (i.e. hormone or barrier method or abstinence) during clinical trial and for a minimum of 12 weeks after the last administration of T601; negative blood pregnancy test for women of childbearing potential (WOCBP) within 7 days before enrollment ;
8. Give informed consent to the study prior to the test and voluntarily sign a written informed consent.

Exclusion Criteria:

1. Received chemotherapy, radiation, biotherapy, endocrine therapy, immunotherapy and other anti-tumor treatments within 4 weeks prior to T601 treatment initiation, except for the following items:

   Received nitrosourea or mitomycin C within 6 weeks before T601 treatment initiation; Orally taken fluorouracil and small-molecule targeted drugs within 2 weeks before T601 treatment initiation or within 5 half-lives of the above drugs (subject to whichever is longer); Received the Chinese medicines with anti-tumor indications within 2 weeks before T601 treatment initiation;
2. Prior participation in another clinical study involving an IMP with last intake within 4 weeks prior to T601 treatment initiation;
3. Received major organ surgery (excluding needle biopsy) or severe trauma within 4 weeks prior to T601 treatment initiation;
4. The adverse reactions of previous anti-tumor therapy have not yet returned to CTCAE 5.0 ≤1 (except the toxicity that the investigator judged as no safety risk, such as hair loss);
5. With clinical symptoms of brain metastasis, spinal cord compression, and cancerous meningitis, or other evidence indicates that the metastasis of the patient's brain and spinal cord has not been controlled, and the investigator judged that the patient was not suitable for inclusion. Patients with clinical symptoms suspected of cerebral or pia mater disease should be excluded by CT/MRI examination;
6. Uncontrolled bacterial, viral or fungal infections requiring systematic treatment;
7. History of immunodeficiency, including positive HIV antibody test;
8. Active chronic hepatitis B (HBV-DNA higher than the lower limit of detection), hepatitis C antibody positive;
9. Patients who are unable to swallow oral drugs;
10. History of serious cardiovascular and cerebrovascular diseases:

    1. Ventricular arrhythmias requiring clinical intervention;
    2. Acute coronary syndrome, congestive heart failure, stroke or other class III or above cardiovascular events within 6 months;
    3. New York Heart Association (NYHA) cardiac function grade ≥II or Left Ventricular Ejection Fraction (LVEF) <50%;
    4. Hypertension uncontrolled by standard treatment;
11. Skin diseases that need systematic treatment;
12. Patients who need long-term use of glucocorticoids (prednisone>10 mg/d or equivalent dose of the same drug) or other immunosuppressive agents during the study period or within 14 days before initiation of T601; Exceptions: local, ocular, intra-articular, intranasal, and inhaled glucocorticoid therapy; Short-term use of glucocorticoids for preventive treatment (e.g. prevention of contrast agent allergy);
13. History of severe systemic reaction or side-effect after vaccinia vaccine injection;
14. Known hypersensitivity to 5-FC or intolerance to 5-FC treatment;
15. Known alcohol or drug dependence;
16. Mental disorders or patients unable or unwilling to comply with the protocol requirements;
17. Pregnant or lactating female patients;
18. Patients who, as determined by the investigator, have other serious systemic diseases or laboratory abnormalities or other reasons, are not eligible to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
AEs (adverse events) | Throughout the whole clinical trial, around 2 years.
  According to NCI CTCAE 5.0., evaluate the AEs and the frequency and severity of adverse events.
Assessment of ORR (objective response rate) | For Part 2, ORR is measured on Day28 for cycle 1, and after cycle 1, ORR is measured when every 2 cycles finished (for Part 2, each cycle is 28 days), until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RECIST v1.1, to assess the ORR of the patients, and to evaluate the efficacy of T601 or T601 in combination with 5-FC
Assessment of ORR (objective response rate) | For Part 3, ORR is measured at the end of each cycle (for Part 3, each cycle is 46 days), until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RECIST v1.1, to assess the ORR of the patients, and to evaluate the efficacy of T601 or T601 in combination with 5-FC
Assessment of ORR (objective response rate) | For Part 4, ORR is measured at the end of each cycle (for Part 4, each cycle is 46 days), until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RECIST v1.1, to assess the ORR of the patients, and to evaluate the efficacy of T601 or T601 in combination with 5-FC
Assessment of DCR (disease control rate) | For Part 2, DCR is measured on Day28 for cycle 1, and after cycle 1, DCR is measured when every 2 cycles finished (for Part 2, each cycle is 28 days), until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RECIST v1.1, to assess the DCR of the patients, and to evaluate the efficacy of T601 or T601 in combination with 5-FC.
Assessment of DCR (disease control rate) | For Part 3, DCR is measured at the end of each cycle (for Part 3, each cycle is 46 days), until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RECIST v1.1, to assess the DCR of the patients, and to evaluate the efficacy of T601 or T601 in combination with 5-FC.
Assessment of DCR (disease control rate) | For Part 4, DCR is measured at the end of each cycle (for Part 4, each cycle is 46 days), until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RECIST v1.1, to assess the DCR of the patients, and to evaluate the efficacy of T601 or T601 in combination with 5-FC.
Assessment of PFS (progression free survival) | For Part 2, PFS is measured on Day28 for cycle 1, and after cycle 1, PFS is measured when every 2 cycles finished (for Part 2, each cycle is 28 days), until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RECIST v1.1, to assess the PFS of the patients, and to evaluate the efficacy of T601 or T601 in combination with 5-FC.
Assessment of PFS (progression free survival) | For Part 3, PFS is measured at the end of each cycle (for Part 3, each cycle is 46 days), until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RECIST v1.1, to assess the PFS of the patients, and to evaluate the efficacy of T601 or T601 in combination with 5-FC.
Assessment of PFS (progression free survival) | For Part 4, PFS is measured at the end of each cycle (for Part 4, each cycle is 46 days), until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RECIST v1.1, to assess the PFS of the patients, and to evaluate the efficacy of T601 or T601 in combination with 5-FC.

SECONDARY OUTCOMES:
Quantification of viral genome in patients' blood samples by Quantitative Polymerase Chain Reaction. | For Part 1, blood samples are collected on Day1, Day4, Day14, Day21 of cycle 1; Day2, Day21 of cycle 2 (for Part 1, each cycle is 21 days).
  to evaluate pharmacokinetics characteristics of T601
Quantification of viral genome in patients' blood samples by Quantitative Polymerase Chain Reaction. | For Part 2, blood samples are collected on Day4, Day14, Day28 of cycle 1.
  to evaluate pharmacokinetics characteristics of T601
Quantification of viral genome in patients' blood samples by Quantitative Polymerase Chain Reaction. | For Part 3, blood samples are collected on Day8, Day15, Day32, Day46 of cycle 1.
  to evaluate pharmacokinetics characteristics of T601
Determination of 5-FC, 5-FU and FBAL concentration in plasma by updated LC/MS/MS method | For Part 2, blood samples are collected on Day7, Day14, Day18 of cycle 1.
  Blood concentration monitoring of 5-FC, 5-FU, FBAL
Determination of 5-FC, 5-FU and FBAL concentration in plasma by updated LC/MS/MS method | For Part 3, blood samples are collected on Day19, Day20 of cycle 1.
  Blood concentration monitoring of 5-FC, 5-FU, FBAL
T601 antibody test by ELISA | For Part 1, Baseline, Day14, Day21 for cycle 1 and Day21 for following cycles (for Part 1, each cycle is 21 days).
  Immunological evaluations
T601 antibody test by ELISA | For Part 2, Baseline, Day14, Day28 for cycle 1 and Day28 for following cycles (for Part 2, each cycle is 28 days).
  Immunological evaluations
T601 antibody test by ELISA | For Part 3, Baseline, Day14, Day32, Day46 for cycle 1 and Day46 for following cycles (for Part 3, each cycle is 46 days).
  Immunological evaluations

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - START-SEH New Drug Phase I Clinical Trial Center, Shanghai